CLINICAL TRIAL: NCT03411850
Title: Disease Modification in Sjogrens Syndrome Measured by Ultrasound: A Pilot Study
Brief Title: Sjogrens Syndrome Measured by Ultrasound
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arthritis & Rheumatism Associates, P.C. (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BMS IM101-560
Record Dates: First submitted 2016-06-30; First posted 2018-01-26 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Abatacept; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orencia (Abatacept) (Active Comparator): Orencia (Abatacept) Intravenous (IV) or Subcutaneous (SQ) injection
  Interventions: Biological: Orencia
- Placebo (Placebo Comparator): Placebo (saline solution) given Intravenous (IV) or Subcutaneous (SQ)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Orencia — FDA approved biologic
  Other Names: Abatacept
  Arms: Orencia (Abatacept)
Other: Placebo
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Ultrasound study focused on salivary gland outcomes in Sjogren's subjects

DETAILED DESCRIPTION:
A 32 week ultrasound study for subject diagnosed with Sjogren's Syndrome. Subjects will receive Orencia (Abatacept) as intervention therapy during this trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with Sjogren's Syndrome

Exclusion Criteria:

* Subjects previously diagnosed with Sarcoidsis
* Subjects with positive for Hepatitis B, Hepatitis C, HIV
* Subjects diagnosed with Cancer within 5 years of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05; Primary Completion 2021-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Salivary gland changes | 32 weeks
  Salivary gland changes detected by ultrasound imaging with elastography

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Rheumatology and Bone Research a division of Arthritis and Rheumatism Associates, P.C., Wheaton, Maryland, United States

IPD SHARING:
Plan to Share IPD: No